CLINICAL TRIAL: NCT02647255
Title: Randomized Trial of Plasma Exchange as Adjunctive Therapy for Severe Crescentic GlomerUlonephritis of IgA NEphropathy (RESCUE Study)
Brief Title: Trial of Plasma Exchange for Severe Crescentic IgA Nephropathy
Acronym: RESCUE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to the rarity and rapid progressive course of the disease, patients were less likely to participate in randomization.
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Hong Zhang, Professor, Principal Investigator, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE
Record Dates: First submitted 2015-12-21; First posted 2016-01-06 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Glomerulonephritis, IGA; Kidney Diseases; Acute Renal Insufficiency; Rapidly Progressive Glomerulonephritis
Keywords: crescentic IgA nephropathy; plasma exchange treatment or plasmapheresis; randomized controlled trial; intensive immunosuppressive treatment; methylprednisolone pulse
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases; Acute Kidney Injury | interventions — Plasma Exchange; Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PE and methylprednisolone pulse (Experimental): Plasma exchange(PE) and methylprednisolone pulse therapy: plasma exchange >7 within 3ws, Volume: 60ml/kg/course; Replacement fluid: 5% albumin or fresh frozen plasma and methylprednisolone pulse therapy Basic treatment: Oral prednisone was tapered from 1 mg/kg/d for 6wks, then diminish 5mg/d every 10d, stop at the sixth month; cyclophosphamide 1.5 mg/kg/d for 3 months, 50mg /d at 3 months and stopped at 6 month.
  Interventions: Procedure: Plasma Exchange (PE); Drug: Methylprednisolone pulse
- Methylprednisolone pulse (Active Comparator): Methylprednisolone pulse alone: methylprednisolone 7-15mg/kg/d 3 times on consecutive or alternate days Basic treatment: Oral prednisone was tapered from 1 mg/kg/d for 6wks, then diminish 5mg/d every 10d, stop at the sixth month; cyclophosphamide 1.5 mg/kg/d for 3 months, 50mg /d at 3 months and stopped at 6 month.
  Interventions: Drug: Methylprednisolone pulse

INTERVENTIONS:
Procedure: Plasma Exchange (PE) — PE treatment>7 within 3weeks; Volume exchanged: 60ml/kg/course; Replacement fluid: 5% Albumin or fresh frozen plasma; PE was performed by dialysis machine (IQ-21, Asahi Japan) and plasma separator (OP- 08W, Asahi Japan)
  Other Names: Plasmapheresis
  Arms: PE and methylprednisolone pulse
Drug: Methylprednisolone pulse — methylprednisolone 7-15mg/kg/d 3 times, Qd. or Qod
  Other Names: Intensive Immunosuppressive treatment

SUMMARY:
Crescentic IgA nephropathy (CreIgAN) has a poor prognosis despite aggressive immunosuppressive therapy. The efficacy of plasma exchange (PE) in CreIgAN is not well defined. This study will evaluate the efficacy and safety of plasma exchange as adjunctive therapy for severe crescentic IgA nephropathy compared to pulse methylprednisolone on a background of oral prednisolone and cyclophosphamide in prevent kidney failure.

DETAILED DESCRIPTION:
IgA nephropathy (IgAN) is one of the most common glomerulonephritides and is characterized by a highly variable clinical course and diverse histopathological lesions. Although most affected individuals develop chronic, slowly progressive renal injury, a subgroup of patients (<5% of all IgAN patients) with diffuse crescent formation, which is termed as crescentic IgA nephropathy (CreIgAN) and often leads to rapidly progressive kidney failure. The recent Kidney Disease: Improving Global Outcomes (KDIGO) guidelines suggest high-dose steroids and cyclophosphamide therapy for CreIgAN. However, this suggestion is mainly based on several small observational studies, and the 1- and 5-year renal survival rates of patients treated with this regimen were as low as 65% and 28%, respectively, in one large cohort of CreIgAN patients. The efficacy of plasma exchange (PE) in severe CreIgAN is not well evaluated, although several anecdotal reports have indicated benefit of PE in combination with immunosuppressive therapies in IgAN patients. Retrospective cohort study in our unite also supported the benefit of PE as additional therapy for CreIgAN patients. However, randomized controlled trial is needed to evaluate the efficacy and safety of plasma exchange as adjunctive therapy for crescentic IgA nephropathy compared to pulse methylprednisolone on a background of oral prednisolone and cyclophosphamide in prevent kidney failure.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven within 3ws
2. Primary IgAN or Henoch-Schönlein Purpura nephritis of crescent >50%(>8 glomeruli)
3. Serum creatinine ≥ 200 μmol/l， rapidly deterioration of renal function

Exclusion Criteria:

1. <14 or >65 years old
2. With high Scr requiring dialysis for≥ 3w
3. Scr>200μmol/L ≥1 yr before entry
4. Main of old crescent ; Fibrous crescent>50%
5. Anti-glomerular basement membrane (GBM) or antineutrophil cytoplasmic antibody (ANCA) antibody positive
6. Women in gestational and lactational period
7. With diabetes or uncontrollable malignant hypertension or Thrombotic Microangiopathy
8. With Malignancy
9. Chronic active infection including HBV hepatitis C virus (HCV) HIV or active tuberculosis
10. Other autoimmune disease
11. A second clearly defined cause of renal failure
12. Contraindication of plasma exchange treatment or steroid pulse
13. Patients who are unlikely to comply with the study protocol in the view of the treating physician.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
End-stage renal disease or death | 12 months after final subject is enrolled
  End-stage renal disease: defined as a need for maintenance dialysis > 6 months; or need kidney transplantation , and death; during follow-up.

SECONDARY OUTCOMES:
Renal remission | 12 months after final subject is enrolled
  Renal remission: defined as the independent of dialysis, or serum creatinine under 200μmol/l within 6 months, and lasts without a first relapse until at least 12 months after randomization
Proteinuria remission | At the 12th month and 36th month after randomization
  Proteinuria remission: defined as proteinuria < 0.5g/d for ≥3months

OTHER OUTCOMES:
Rate of serious adverse events | From 12 months after first subject enrolled to 12 months after final subject is enrolled
  Serious adverse events are defined as:
  Clinically apparent gastrointestinal haemorrhage requiring hospitalization or prolonging the time of hospitalization.
  Serious infections requiring hospitalization or prolonging the time of hospitalization.
  Severe allergic reaction requiring hospitalization or prolonging the time of hospitalization.
  Chronic viral infection, including HIV hepatitis B virus(HBV) and HCV Other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, MD, PHD, Study Director — Renal Division, Department of Medicine, Peking University First Hospital;Peking University Institute of Nephrology
Locations (2):
- China (2):
  - Renal Division, Department of Medicine, Peking University First Hospital, Beijing, Beijing Municipality
  - Renal division, Peking University First Hospital, Beijing, Beijing Municipality

REFERENCES:
- [Background] Suzuki H, Kiryluk K, Novak J, Moldoveanu Z, Herr AB, Renfrow MB, Wyatt RJ, Scolari F, Mestecky J, Gharavi AG, Julian BA. The pathophysiology of IgA nephropathy. J Am Soc Nephrol. 2011 Oct;22(10):1795-803. doi: 10.1681/ASN.2011050464. Epub 2011 Sep 23. PMID 21949093
- [Background] Lv J, Yang Y, Zhang H, Chen W, Pan X, Guo Z, Wang C, Li S, Zhang J, Zhang J, Liu L, Shi S, Wang S, Chen M, Cui Z, Chen N, Yu X, Zhao M, Wang H. Prediction of outcomes in crescentic IgA nephropathy in a multicenter cohort study. J Am Soc Nephrol. 2013 Dec;24(12):2118-25. doi: 10.1681/ASN.2012101017. Epub 2013 Sep 12. PMID 24029421
- [Background] Abe T, Kida H, Yoshimura M, Yokoyama H, Koshino Y, Tomosugi N, Hattori N. Participation of extracapillary lesions (ECL) in progression of IgA nephropathy. Clin Nephrol. 1986 Jan;25(1):37-41. PMID 3955907
- [Background] Tang Z, Wu Y, Wang QW, Yu YS, Hu WX, Yao XD, Chen HP, Liu ZH, Li LS. Idiopathic IgA nephropathy with diffuse crescent formation. Am J Nephrol. 2002 Sep-Dec;22(5-6):480-6. doi: 10.1159/000065281. PMID 12381947
- [Background] Tumlin JA, Lohavichan V, Hennigar R. Crescentic, proliferative IgA nephropathy: clinical and histological response to methylprednisolone and intravenous cyclophosphamide. Nephrol Dial Transplant. 2003 Jul;18(7):1321-9. doi: 10.1093/ndt/gfg081. PMID 12808169
- [Background] Pankhurst T, Lepenies J, Nightingale P, Howie AJ, Adu D, Harper L. Vasculitic IgA nephropathy: prognosis and outcome. Nephron Clin Pract. 2009;112(1):c16-24. doi: 10.1159/000210570. Epub 2009 Apr 3. PMID 19342865
- [Background] Jayne DR, Gaskin G, Rasmussen N, Abramowicz D, Ferrario F, Guillevin L, Mirapeix E, Savage CO, Sinico RA, Stegeman CA, Westman KW, van der Woude FJ, de Lind van Wijngaarden RA, Pusey CD; European Vasculitis Study Group. Randomized trial of plasma exchange or high-dosage methylprednisolone as adjunctive therapy for severe renal vasculitis. J Am Soc Nephrol. 2007 Jul;18(7):2180-8. doi: 10.1681/ASN.2007010090. Epub 2007 Jun 20. PMID 17582159
- [Background] Nicholls K, Becker G, Walker R, Wright C, Kincaid-Smith P. Plasma exchange in progressive IgA nephropathy. J Clin Apher. 1990;5(3):128-32. doi: 10.1002/jca.2920050303. PMID 2345159
- [Background] Lai KN, Lai FM, Leung AC, Ho CP, Vallance-Owen J. Plasma exchange in patients with rapidly progressive idiopathic IgA nephropathy: a report of two cases and review of literature. Am J Kidney Dis. 1987 Jul;10(1):66-70. doi: 10.1016/s0272-6386(87)80014-8. PMID 3300287
- [Background] Fujinaga S, Ohtomo Y, Umino D, Mochizuki H, Murakami H, Shimizu T, Yamashiro Y, Kaneko K. Plasma exchange combined with immunosuppressive treatment in a child with rapidly progressive IgA nephropathy. Pediatr Nephrol. 2007 Jun;22(6):899-902. doi: 10.1007/s00467-006-0428-4. Epub 2007 Feb 7. PMID 17285293
- [Background] Nicholls K, Walker RG, Dowling JP, Kincaid-Smith P. "Malignant" IgA nephropathy. Am J Kidney Dis. 1985 Jan;5(1):42-6. doi: 10.1016/s0272-6386(85)80134-7. PMID 3966468
- [Background] Roccatello D, Ferro M, Coppo R, Giraudo G, Quattrocchio G, Piccoli G. Report on intensive treatment of extracapillary glomerulonephritis with focus on crescentic IgA nephropathy. Nephrol Dial Transplant. 1995 Nov;10(11):2054-9. PMID 8643167
- [Background] Schwartz J, Winters JL, Padmanabhan A, Balogun RA, Delaney M, Linenberger ML, Szczepiorkowski ZM, Williams ME, Wu Y, Shaz BH. Guidelines on the use of therapeutic apheresis in clinical practice-evidence-based approach from the Writing Committee of the American Society for Apheresis: the sixth special issue. J Clin Apher. 2013 Jul;28(3):145-284. doi: 10.1002/jca.21276. PMID 23868759
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- See also: KDIGO Clinical Practice Guideline for Glomerulonephritis (GN) — http://kdigo.org/home/glomerulonephritis-gn/